CLINICAL TRIAL: NCT06304701
Title: Analysis on Graphic Tablet of Motor and Cognitive Components of Written Production in Adults With and Without Autism Spectrum Disorder
Brief Title: Handwritten Text Production in Adults With Autism
Acronym: PEMTAA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier de Niort (Other)
Collaborators: University of Poitiers (Other)
Responsible Party: Principal Investigator, Evan Launay, Psychologist and PhD student, Centre Hospitalier de Niort
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI-2023-08
Record Dates: First submitted 2024-02-12; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Autism Spectrum Disorder
Keywords: Written production; Handwriting; Graphomotor skills; Language; Graphic tablet
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Intervention Model Description: The study is part of category 2 of research involving humans and which corresponds to an interventional study with minimal risks and constraints. The patient is asked to return to carry out this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm : Adults with autism spectrum disorder (Experimental): All of the interventions described below
  Interventions: Diagnostic Test: Cognitive and writing tests
- Control arm : Adults with typical development (Active Comparator): All of the interventions described below
  Interventions: Diagnostic Test: Cognitive and writing tests

INTERVENTIONS:
Diagnostic Test: Cognitive and writing tests — * Wechsler Adult Intelligence Scale - fourth edition (Similarities and Vocabulary subtests)
  * MASC (Movie for assessment of social cognition)
  * Rey figure
  * BHK (Quick Writing Assessment Scale)
  * Descriptive text writing
  * Persuasive text writing

SUMMARY:
The main objective is to assess the psycholinguistic and graphomotor characteristics of written production in patients with ASD.

The secondary objectives are:

* Identifying links between specific deficits of ASD and difficulties in written production.
* Identifying links between the severity of ASD and difficulties in written production.

The primary evaluation criterion is the quantity of written production, namely the number of words produced in 5 minutes on a text copying task (BHK) and in 15 minutes on each of the two written production tasks (descriptive and persuasive).

The secondary evaluation criteria are:

* Graphomotor indicators of written production (writing speed, pre-writing time, pause time, writing time, handwriting size, results obtained in BHK (number of words produced, letter height, line parallelism, telescoping, ambiguous letters).
* Cognitive and psycholinguistic indicators of written production (presence of titles, presence of paragraphs, number of sentences, number of words per sentence, lexical richness, lexical field, number of action verbs, morphological complexity, number of syntactic markers related to oneself, number of syntactic markers related to others, number of spelling errors, evaluation of the overall quality of the produced text).
* Results obtained in tests (writing habits questionnaire, Autism Diagnostic Observation Scale (second edition), Wechsler Adult Intelligence Scale (fourth edition) - Similarities subtest, Wechsler Adult Intelligence Scale (fourth edition) - Vocabulary subtest, Rey Figure, MASC).

DETAILED DESCRIPTION:
Context :

Autism Spectrum Disorder (ASD) is one of the neurodevelopmental disorders (NDD) characterized by persistent deficits in communication and social interaction, and restricted and repetitive patterns of behavior, interests, and activities (DSM-5 diagnostic criteria; American Psychiatric Association, 2013). These symptoms are present from early developmental stages and correspond to neurological conditions characterized by structural and/or functional brain abnormalities.

While diagnosis is typically made in childhood (average age of 4 years (Rogé, 2019)), many adults seek diagnostic evaluation for ASD from autism resource centers (CRA). This is partly due to the diversity of symptoms that can lead to a 'diagnostic odyssey' spanning several years (Rutherford et al., 2016). Even though the dyad identified by DSM-5 allows for precise diagnosis, many other clinical signs can be found in patients with ASD (mood disorders, sleep disorders, impulsivity/hyperactivity, anxiety, motor disorders, language disorders, etc.), which can complicate diagnosis and delay the implementation of early and appropriate intervention.

In this context, an interesting avenue is the study of writing characteristics in patients with ASD. Indeed, several studies show that patients with ASD present deficits in motor skills as well as in several psycholinguistic domains such as grammar, morphology, and phonology (Habib et al., 2019). Furthermore, individuals with ASD may exhibit specific semantic and pragmatic impairments (Bishop, 1989). These findings may provide additional useful clues in a perspective of differential diagnosis and understanding of cognitive functioning.

ELIGIBILITY:
Inclusion Criteria for experimental group only:

* ASD diagnosis according to DSM-5 criteria and established by an interdisciplinary

Inclusion Criteria for both experimental and control groups:

* Age ≥ 18 years Age ≥ 18 years and matching typical adult subjects to ASD individuals in age (plus or minus 5 years), sex, and education level
* The person participating in the research has read, understood, and signed the study consent form
* The person is proficient in the French language
* The person is affiliated with a social security system

Exclusion Criteria for experimental group only:

* Diagnosis of any other NDD than ASD (e.g., Attention Deficit Hyperactivity Disorder, Specific Learning Disorder, Language Disorder, Coordination Disorder, Intellectual Disorder)

Exclusion Criteria for control group only:

- Diagnosis of any NDD (ASD, Attention Deficit Hyperactivity Disorder, Specific Learning Disorder, Language Disorder, Coordination Disorder, Intellectual Disorder)

Exclusion Criteria for both experimental and control groups:

* Refusal of the individual to participate in the study
* Presence of severe visual impairment
* Known pregnancy
* Individual deprived of liberty
* Individual under guardianship or curators
* Presence of concurrent psychotropic medication treatments not stabilized, initiated within the last 2 months: antipsychotics, mood stabilizers, antiepileptics, psychostimulants, antidepressants
* Presence of upper limb motor impairment, with or without devices
* Presence of diagnosed neurological or psychiatric disorders (e.g., Schizophrenia Spectrum Disorder or other psychotic disorders), presence of a general or metabolic pathology known to have an impact on cognitive efficiency and/or motor skills of the individual (e.g., Epilepsy, Tics and Tourette Syndrome, Neuro-muscular Syndrome, Metabolic Neurological Syndromes, neoplasms)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-29 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Assessment of psycholinguistic and graphomotor characteristics of written production in patients with autism spectrum disorder (asd) | 18 months
  Number of words produced in both 3 written production tasks (copy, descriptive text, and persuasive text) : adults with ASD vs adults with typical development

SECONDARY OUTCOMES:
Identifying links between specific deficits of ASD and difficulties in written production | 18 months
  Identifying links between theory of mind (MASC results), which is one of the main explicative model of the autistic functioning, and number of words produced in both 3 written production tasks. Indeed, the writing activity involves taking into account the recipient, and thus the theory of mind.
Identifying links between the severity of ASD and difficulties in written production | 18 months
  Identifying links between the severity of ASD (ADOS-2 results) and number of words produced in both 3 written production tasks. Indeed, the severity of ASD can affect the ability to communicate, which is one of the diagnostic criteria of ASD, and thus the ability to produce a text.

CONTACTS AND LOCATIONS:
Overall Officials: Evan E Launay, Mr, Principal Investigator — Hospital Center of Niort (France)
Locations (1):
- Centre Hospitalier de Niort, Niort, France

IPD SHARING:
Plan to Share IPD: No